CLINICAL TRIAL: NCT07082933
Title: Long-term Survival and Influencing Factors of Patients With Pulmonary Arterial Hypertension and diabetes-a Multicenter Retrospective Cohort Study
Brief Title: Long-term Survival and Influencing Factors of Patients With Pulmonary Arterial Hypertension and Diabetes
Status: Not yet recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY-20252240
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
Keywords: Pulmonary arterial hypertension; Diabetes; Mortality
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pulmonary arterial hypertension combined with diabetes: patients with pulmonary arterial hypertension and diabetes
  Interventions: Other: Standard medical treatment
- pulmonary arterial hypertension without comorbid diabetes: pulmonary arterial hypertension without comorbid diabetes
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Other: Standard medical treatment — Standard medical treatment

SUMMARY:
This is a multicenter retrospective cohort study on pulmonary arterial hypertension. It is expected to collect data from no less than 5,000 patients to compare the long-term overall survival of patients with and without diabetes, and analysis the risk factors of the overall survival .

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 to 80 years with full capacity for civil conduct.
* Patients diagnosed with pulmonary hypertension by community-level and/or higher-level medical institutions.

Exclusion Criteria:

* Patients with malignant tumors.
* Other physical conditions judged by the researchers as making the patients ineligible to participate in the clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with pulmonary hypertension
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 10 years
  Time from diagnosis of pulmonary hypertension to death

SECONDARY OUTCOMES:
Pulmonary Artery Pressure(PAP) | baseline

OTHER OUTCOMES:
Brain natriuretic peptide | baseline
blood glucose | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Yue Zhang, Doctor, Principal Investigator — Department of Health Management, Xijing Hospital, Air Force Medical University

IPD SHARING:
Plan to Share IPD: No